CLINICAL TRIAL: NCT01330446
Title: Armodafinil for Persistent Patient-Reported Fatigue Following Radiation Therapy for Head and Neck Cancer: a Randomized Phase II Study
Brief Title: Single Agent Armodafinil for Patient-Reported Fatigue Following Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-0557; R01 026582-26 (Other Grant/Funding Number: National Cancer Institute); NCI-2011-00881 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Head And Neck Cancer; Fatigue
Keywords: Head and Neck Cancer; HNC; Fatigue; Patient-Reported Fatigue; Fatigue-Symptom Intervention; Postoperative Radiation Therapy; Postoperative Chemoradiation Therapy; Armodafinil; Nuvigil; Placebo; Sugar Pill; Questionnaires; Surveys
MeSH Terms: conditions — Head and Neck Neoplasms; Fatigue | interventions — Modafinil; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Armodafinil (Experimental): 50 mg the first 3 days, 100 mg the next 4 days, and 150 mg for the remaining treatment period.
  Interventions: Drug: Armodafinil; Behavioral: Questionnaires
- Placebo (Placebo Comparator): 1 Placebo by mouth every morning for a 28 day cycle.
  Interventions: Other: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Armodafinil — 50 mg the first 3 days, 100 mg the next 4 days, and 150 mg for the remaining treatment period.
  Other Names: Nuvigil
  Arms: Armodafinil
Other: Placebo — 1 by mouth every morning for a 28 day cycle.
  Other Names: Sugar Pill
  Arms: Placebo
Behavioral: Questionnaires — Series of questionnaires completed at different time points before, during, and at study completion.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if armodafinil can reduce fatigue and other common symptoms in patients that have received treatment for head and neck cancer.

DETAILED DESCRIPTION:
Armodafinil is designed to stimulate the central nervous system, which may increase wakefulness and reduce fatigue.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

Study Groups:

If participant is found eligible to take part in this study, participant will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Group 1 will take armodafinil. Group 2 will take a placebo. A placebo is a substance that looks like the study drug but has no active ingredients.

Neither participant nor the study staff will know if participant is receiving the study drug or the placebo. However, if needed for participant's safety, the study staff will be able to find out what participant is receiving.

Study Drug Administration:

Participant will take the study drug/placebo every day for 4 weeks starting the morning after participant has enrolled in this study. Participant will take the study drug/placebo in the morning with a full glass (8 ounces) of water. Participant may take the study drug/placebo with or without food. If the dose causes an upset stomach, participant should take it with food. If participant has trouble swallowing the dose of study drug/placebo, the study staff will tell participant of different ways of taking it. Participant will be given a pamphlet with more information about how to take the study drug/placebo.

Symptom Questionnaires:

Before participant starts taking the study drug/placebo, the following tests and procedures will be performed:

°Participant will complete 6 questionnaires about participant's fatigue, sleepiness, and other symptoms as well as participant's quality of life and participant's ability to work. These questionnaires should take about 20 minutes to complete total.

Throughout the study, participant will complete 2 of the symptom questionnaires listed above 2 times every week while participant is on study, including during the Open-label Extension Phase (described below). Participant may complete the questionnaires over the phone using the Interactive Voice Response (IVR) system or with a member of the study staff. Another option is to complete the questionnaires during a routinely scheduled visit outside of this study. If participant completes the questionnaires over the phone, the study staff or the IVR system will call participant at a time that is convenient for participant. If the questionnaires are completed through the IVR system, the study staff will give participant the information participant needs to report participant's symptoms by using the system. If the questionnaires are completed with the study staff, she/he will ask participant the questions and record participant's answers on paper or enter them into a computer.

When participant completes the questionnaires for the second time each week, participant will also be asked if participant is taking participant's study drug/placebo as instructed and participant will be asked about any side effects participant may be having. If the questionnaires were completed through the IVR system, the study staff will contact participant and ask participant if participant is taking participant's study drug/placebo as instructed and about any side effects participant may be having.

At the end of Week 4, participant will complete the same set of 6 questionnaires that participant completed at the beginning of the study. Participant will also complete a questionnaire about participant's thoughts on the study drug/placebo. Participant will also be asked about any changes in drugs (both prescribed and over the counter) that participant may be taking. This should take about 30 minutes.

Open-label Extension:

At the end of Week 4, if participant was in Group 1 and participant did not have any intolerable side effects, participant will be able to continue taking armodafinil for an additional 4 weeks. If participant was in Group 2 and participant did not have any intolerable side effects, participant will be given the option to begin receiving armodafinil for 4 weeks.

No matter what participant chooses, participant will not be told whether participant was taking the study drug or the placebo during the first 4 weeks of the study.

If participant is in the open-label extension phase, at the end of Week 8, participant will complete the same set of 6 questionnaires that participant completed at the beginning of the study. Participant will also complete a questionnaire about participant's thoughts on the study drug/placebo. This should take about 30 minutes.

Length of Treatment:

Participant will receive the study drug/placebo for either 4 or 8 weeks. Participant will be taken off study if intolerable side effects occur or if the study doctor thinks it is in participant's best interest.

Follow-Up:

After participant's last dose of the study drug/placebo, participant will continue to complete 2 symptom questionnaires for another 4 weeks. The last time participant completes the 2 questionnaires, participant will complete an additional 3 questionnaires that participant completed at the beginning of the study.

Additional Information:

Any information about the side effects participant may have that are collected during this study will not be reported to participant's regular doctor. Participant should tell participant's regular doctor about all symptoms and/or side effects that participant had. Participant will given a hot line phone number to call the study staff if participant has any side effects from the study drug/placebo.

Another option to complete the questionnaires at Weeks 4, 8, and 12 is to receive questionnaire packets during the baseline assessment and to mail them back to the study coordinator. The study staff will contact participant to remind participant when it is time to complete them.

This is an investigational study. Armodafinil is FDA-approved and commercially available to treat narcolepsy (falling asleep at unexpected times), obstructive sleep apnea, and shift work sleep disorder. It is also FDA-approved and commercially available to treat sleepiness in patients with excessive sleepiness. Its use in this study is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were treated with either definitive or postoperative radiation or chemoradiation therapy for HNC with moderate to severe levels of patient reported fatigue, at 6 or more weeks after completing all planned cancer therapy. Patients who rated their fatigue level at 5 or greater on a 0 to 10 scale during any follow-up clinic visits at MD Anderson.
2. Male and female patients >= 18 years old.
3. Patients who speak English (due to the novel research and its complexity, we are only accruing English-speaking patients to the protocol).
4. Patients must agree to discontinue any current herbal supplement use, and refrain from taking any herbal supplement while on protocol.
5. Patients must be willing and able to review and understand informed consent documents and to provide written consent.
6. Women of childbearing potential (women who are not postmenopausal for at least 1 year and are not surgically sterile) must have a negative urine pregnancy test.
7. Sexually active males and females must agree to use effective birth control or to be abstinent for the duration of the study period.
8. Women currently taking birth control pills or planning to start birth control pills must agree to an additional method of birth control (either abstinence or a barrier method) while on the study medication and for 1 additional month after study completion.

Exclusion Criteria:

1. Patients who rated their fatigue level at 4 or less over the past 24 hours based on the fatigue at its worst item of the BFI.
2. Patients with clinical evidence of active persistent cancer or progressive disease after completing planned cancer therapy, or with active recurrent cancer.
3. Patients with potential medical or other underlying causes of fatigue, as determined by the treating physician or PI
4. Patients with Hb <10.5 g/dL within previous 2 weeks.
5. Patients with untreated or uncontrolled hypothyroidism, or TSH > ULN or free T4 < lower level of normal within previous 2 weeks.
6. Patients with underlying cardiac or pulmonary disease resulting in dyspnea, hypoxia, or hypercapnia.
7. Patients with a Karnofsky performance status <70
8. Patients less than 18 years old
9. Patients who are enrolled and receiving active treatment in other symptom intervention trials or who are in the treatment phase of another clinical trial
10. Patients with pre-existing psychosis or bipolar disorder
11. Patients with pre-existing renal impairment, as evidenced by serum creatinine > ULN on the most recent blood work, done at least within the previous 2 weeks.
12. Patients with pre-existing cirrhosis or hepatic impairment or with abnormal liver function test as evidenced by total bilirubin > 1.5 x ULN or 2 times the upper limit of normal of alkaline phosphatase (ALP), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) on the most recent blood work, done at least within the previous 2 weeks.
13. Patients with pre-existing Tourette's syndrome
14. Patients who have used monoamine oxidase (MAO inhibitors) within the past 14 days
15. Patients undergoing abrupt discontinuation of ethanol or sedatives (including benzodiazepines)
16. Patients currently taking, or having taken within the previous 1 month, armodafinil, modafinil, amphetamine, or methylphenidate
17. Patients on anticoagulants (i.e. warfarin, coumadin, or heparin) or clopidogrel
18. Patients with a history of clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reactions
19. Patients with a history of angina or cardiac ischemia, a recent history of myocardial infarction (within the past 1 year) or left ventricular hypertrophy, or patients with mitral valve prolapse
20. Patients with uncontrolled hypertension or tachycardia, as determined by treating physician
21. Patients who are pregnant, breastfeeding, or planning to become pregnant during the study period and for 1 month after stopping the study drug.
22. Female patients who are currently on birth control pills as primary means of contraception, but are not willing to seek an additional effective method of contraception (such as barrier method) during the study period and for 1 month after stopping the study drug.
23. Patients with a history of CNS stimulant abuse, such as methylphenidate, dextroamphetamine, or modafinil.
24. Patients with major depressive disorder or severe depression (a score of 13 or greater on the BDI Fast Screen (BDI-FS). If this is the case, we will notify their treating physician for appropriate management or referral.
25. Patients with current or a history of suicidal ideation.
26. Patients currently taking midazolam, cyclosporine, ethinyl estradiol, or triazolam
27. Patients currently taking carbamazepine, phenobarbital, rifampin, aminoglutethimide, nafcillin, nevirapine, phenytoin, azole antifungals, clarithromycin, diclofenac, doxycycline, erythromycin, imatinib, isoniazid, nefazodone, nicardipine, propofol, protease inhibitors, quinidine, telithromycin, or verapamil
28. Patients currently taking omeprazole, diazepam, propanolol, chlomipramine (or other tricyclic antidepressants), citalopram, methsuximide, or sertraline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05-19 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary B. Gunn, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.utmdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Armodafinil; Placebo: 50 mg the first 3 days, 100 mg the next 4 days, and 150 mg for the remaining treatment period. By mouth every morning for a 28 day cycle.
Period: Overall Study
Arm/Group | Armodafinil | Placebo
Started | 13 | 13
Completed | 8 | 9
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Brief Fatigue Inventory-Worst
Description: The primary outcome measure is item 3 on the Brief Fatigue Inventory (BFI) scale: "Please rate your fatigue (weariness, tiredness) by circling the one number that best describes your WORST level of fatigue during past 24 hours." The item is on a 10-point Likert scale from 0 (no fatigue) to 10 (as bad as you can imagine). Thus, higher values represent worse outcomes. The primary outcome measure is the area under the curve (AUC), using the trapezoidal rule, for the BFI-Worst Fatigue scores over 28 days. The range for BFI-Worst Fatigue AUC is from 0 to 280.
Time Frame: 4-6 weeks
Population: The primary outcome measure is an item on a scale, i.e., has no units, the AUC also has no units.
Measure: Median (Full Range); unit: scores on a scale*day
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 12
scores on a scale*day | 166.8 [70.5 to 243.0] | 154.8 [79.0 to 209.0]

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Armodafinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/13 | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil (N=13) | Placebo (N=13)
Insomnia (Psychiatric disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2
Mania (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT01330446/Prot_SAP_000.pdf